CLINICAL TRIAL: NCT01724190
Title: Effect of Vitamin D Supplementation on Rate of Partial Clinical Remission in Children and Adolescents With Type 1 Diabetes
Brief Title: Effect of Vitamin D on the Honeymoon Period in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathryn Obrynba, Endocrinology Fellow, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 285412
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Vitamin D; Clinical Remission
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Subjects will receive oral vitamin D supplementation, 3000 IU daily over the course of 9 months.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Subjects will receive a placebo solution daily over the course of 9 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D
  Other Names: Cholecalciferol
  Arms: Vitamin D
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if supplementation with Vitamin D in children and adolescents with newly diagnosed type 1 diabetes increases the number of patients who enter the honeymoon period.

DETAILED DESCRIPTION:
Type 1 diabetes is an autoimmune disease characterized by destruction of the insulin secreting beta-cells of the pancreas. There is evidence that Vitamin D may play a role in the initial risk of development of autoimmune disease, including type 1 diabetes. However, Vitamin D may also play a role the natural progression of type 1 diabetes by altering innate insulin secretion and sensitivity and by influencing systemic inflammation, directly at the level of the beta-cell. Studies have shown that Vitamin D insufficiency or deficiency is frequently reported in children and adolescents with type 1 diabetes. A majority of newly diagnosed patients with type 1 diabetes enter a period of partial clinical remission, characterized by low or even absent insulin requirements, also known as a honeymoon period. This honeymoon period is associated with improved metabolic control, near normal insulin sensitivity, and recovery of beta-cell function leading to preservation of endogenous insulin secretion. We hypothesize that supplementation with Vitamin D in children and adolescents with newly diagnosed type 1 diabetes will halt the destructive process within the beta cell and improve beta-cell function by increasing endogenous insulin secretion and decreasing systemic inflammation, thereby increasing the rate of partial clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents ages 4-18 years old with newly diagnosed type 1 diabetes.

Exclusion Criteria:

* age less than 4 years
* pregnant females
* previous or known history of Vitamin D deficiency or insufficiency
* current use of Vitamin D supplementation or multi-vitamin containing >800 IU daily
* or concurrent development and/or history of other significant systemic illness or non-endocrine autoimmune disorder.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Stephens, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Subjects will receive oral vitamin D supplementation, 3000 IU daily over the course of 9 months.
  Vitamin D
- Placebo: Subjects will receive a placebo solution daily over the course of 9 months.
  Placebo
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 19 | 18
Completed | 15 | 14
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 14 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.875 (2.59) | 11.6 (3.28) | 10.7 (3.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: IDAA1c
Description: Our primary outcome measure will be to determine the rate of partial clinical remission at 9 months of disease duration, which will be assessed by determining insulin dose adjusted hemoglobin A1c (IDAA1c) using the formula (HbA1c% + [4 x insulin dose u/kg/day]). A IDAA1c <9 will be indicative of partial clinical remission.
Time Frame: 9 months disease duration
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 15 | 14
Participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes